CLINICAL TRIAL: NCT00986999
Title: Pilot Study of the Effect of Low-Dose Rosuvastatin on Endothelial Function, Oxidative Stress and Inflammatory Parameters in HIV-Infected Individuals With Low HDL Cholesterol Levels and Low to Normal LDL Cholesterol Levels
Brief Title: Effect of Rosuvastatin on Endothelial Function
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: poor enrollment
Sponsor: University of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H002; R01HL095135 (NIH)
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Results first posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: HIV Infections; Cardiovascular Disease
Keywords: HIV infected; treatment experienced
MeSH Terms: conditions — HIV Infections; Cardiovascular Diseases | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rosuvastatin (Experimental): rosuvastatin 10 mg qd increased to 20 mg qd as tolerated
  Interventions: Drug: rosuvastatin

INTERVENTIONS:
Drug: rosuvastatin — rosuvastatin 20 mg tablet, 1/2 tab qd increased to a full tablet qd as tolerated x 6 months with optional extension to 2 years
  Other Names: Crestor

SUMMARY:
Rosuvastatin belongs to a class of medications commonly called "statins" which are medications given for high low density lipoprotein (LDL) 'bad' cholesterol to prevent atherosclerosis (hardening of blood vessels) and lower risk of heart attacks and other circulation problems. Recent studies in the general non-HIV infected population have shown that the beneficial effect of statins in preventing circulation problems is larger than would be expected from lowering of LDL-cholesterol alone. It has been suggested that the additional beneficial effect of statins may be due to the anti-inflammatory effect of statins.

The risk of heart attacks and other circulation problems may be high in HIV infected individuals. This may be due to the inflammatory stress effects of HIV. The main purpose of the study is to see if rosuvastatin will have a beneficial effect on the circulatory system in HIV infected individuals even in those who do not have high LDL cholesterol levels. Therefore, in HIV-infected individuals with normal or low LDL cholesterol levels but with evidence of low HDL cholesterol levels which may be a sign of low grade inflammation, the study will look at whether 3 months of rosuvastatin will lead to improvement in brachial artery flow-mediated dilatation (FMD), a marker of early atherosclerosis (hardening of the blood vessels).

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Age > 18 years old
* On stable antiretroviral therapy for > 6 months with no plans to change therapy during the treatment phase of the study
* Plasma HIV RNA < 50 copies/mL
* Karnofsky performance score > 70 within 30 days prior to study entry
* Ability to understand and sign informed consent
* Following laboratory values obtained within 30 days prior to randomization:

  * Absolute neutrophil count (ANC) > 750/mm3
  * Hemoglobin >/= 8.0 g/dL
  * Platelets >/= 50,000/mm3
  * ALT (SGPT) and AST (SGOT) < 2.5 x ULN
  * Fasting glucose < 126 mg/dL
  * TSH < 3.0 mIU/L
* HDL-C < 50 mg/dL in men, < 55 mg/dL in women
* Direct LDL-C </= 130 mg/dL
* Calculated creatinine clearance > 50 mL/min
* Willing to be treated with rosuvastatin or be on an observational arm for a minimum of 3 months
* Female subject must not participate in a conception process (active attempt to become pregnant) or be post-menopausal. If participating in sexual activity that could lead to pregnancy, the subject must use contraception while receiving study medication and 30 days after stopping the medication

Exclusion criteria

* History of past cardiovascular event
* Acute illnesses or active AIDS-defining opportunistic infection (OI) within 30 days prior to entry
* Other chronic illness including diabetes, autoimmune diseases, and endocrinopathies
* Serology positive for hepatitis B surface antigen or hepatitis C antibody
* Signs and symptoms of liver failure
* Receipt of supraphysiologic glucocorticoid therapy within 3 months prior to study entry
* Use of lipid lowering agents within 30 days prior to study entry
* Receipt of an HIV vaccine or investigational agents
* Pregnancy or breast-feeding
* Presence of any active malignancy within the last 5 years
* Severe Hypertension (Systolic >/= 180 or Diastolic >/= 110 mm Hg)
* Use of oral postmenopausal hormone replacement therapy
* Known hypersensitivity to rosuvastatin
* Active drug or alcohol dependence
* Any acute illness within 30 days prior to study entry that, in the opinion of the site investigator, would interfere with participation in the study.
* Use of lopinavir/ritonavir (Kaletra) as part of current HIV antiretroviral regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-09; Primary Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Shikuma, MD, Principal Investigator — Hawaii Center for AIDS, John A. Burns School of Medicine, University of Hawaii
Locations (1):
- Hawaii Center for AIDS, Honolulu, Hawaii, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rosuvastatin
Started | 7
Completed | 6
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Flow Mediated Dilatation (FMD) of the Brachial Artery
Time Frame: 3 months
Population: Not analyzed
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in HIV Biomarkers of Immune Activation to Include CD38 and CD69 Expression on T Cells and CD16 and CD69 Expression on Monocytes
Time Frame: 3 months
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Mitochondrial-specific Oxidative Stress (Mt-specific 8-oxo-dG) and Oxidative Phosphorylation (OXPHOS) Protein/Enzyme Activity [Complex I and Complex IV] Levels
Time Frame: 3 months
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Glucose Homeostasis and Insulin Resistance as Assessed by Oral Glucose Tolerance Testing
Time Frame: 3 months
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Total, HDL and LDL Cholesterol and Triglyceride Levels
Time Frame: 3 months
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in hsCRP
Time Frame: 3 months
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Rosuvastatin
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes